CLINICAL TRIAL: NCT00024414
Title: Phase II Open-Label Study of Taxoprexin (DHA-Paclitaxel) Injection by 2-Hour Intravenous Infusion in Patients With Metastatic Hormone-Refractory Prostate Cancer
Brief Title: DHA-Paclitaxel in Treating Patients With Metastatic Prostate Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Theradex (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068930; THERADEX-P01-00-04; JHOC-01011003; PROTARGA-P01-00-04
Record Dates: First submitted 2001-09-13; First posted 2003-01-27 (Estimated); Last update posted 2008-07-24 (Estimated); Status verified 2003-03

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — docosahexaenoyl-paclitaxel

INTERVENTIONS:
Drug: DHA-paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of DHA-paclitaxel in treating patients who have metastatic prostate cancer that has not responded to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the objective tumor response rate or prostate-specific antigen response, duration of response, and time to disease progression in patients with metastatic hormone-refractory prostate cancer treated with DHA-paclitaxel.
* Determine the overall survival of patients treated with this drug.
* Determine the toxicity profile of this drug in these patients.
* Assess the quality of life of patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive DHA-paclitaxel IV over 2 hours on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, every 2 courses, and off study.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 18-50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the prostate

  * Progressive metastatic disease on continuous hormonal therapy (e.g., orchiectomy or luteinizing hormone-releasing hormone (LHRH) agonist)
  * Progressive disease is defined by all of the following:

    * Measurable disease or lesions on bone scan
    * Increases in prostate-specific antigen (PSA) levels on at least 2 consecutive measurements
    * Continued PSA elevation after cessation of prior antiandrogen therapy (4 weeks after flutamide and nilutamide and 8 weeks after bicalutamide)
* PSA level at least 5 ng/mL
* Serum testosterone level less than 50 ng/mL

  * Patients who have not undergone prior surgical castration should continue primary androgen suppression (LHRH agonist)
* No known or clinical evidence of CNS metastasis

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT or SGPT no greater than 2.5 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN

Cardiovascular:

* No uncontrolled ventricular arrhythmia
* No myocardial infarction within the past 3 months
* No superior vena cava syndrome

Neurologic:

* No peripheral neuropathy greater than grade 1
* No uncontrolled major seizure disorder
* No spinal cord compression

Other:

* No psychiatric disorder that would preclude informed consent
* No unstable or serious concurrent medical condition
* No concurrent serious infection requiring parenteral therapy
* No other prior or concurrent malignancy except:

  * Curatively treated nonmelanoma skin cancer OR
  * Other cancer curatively treated with surgery alone that has not recurred for more than 5 years
* Fertile patients must use effective contraception during and for at least 6 months after study therapy

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent immunotherapy

Chemotherapy:

* No prior taxanes
* Prior mitoxantrone or prednisone for metastatic disease allowed
* At least 28 days since prior chemotherapy and recovered
* No other concurrent chemotherapy

Endocrine therapy:

* See Disease Characteristics
* No concurrent hormonal therapy

Radiotherapy:

* No prior samarium SM 153 lexidronam pentasodium or strontium chloride Sr 89
* Prior external radiotherapy for metastatic disease allowed
* At least 28 days since prior large-field radiotherapy and recovered
* No concurrent radiotherapy, including whole-brain radiotherapy for documented CNS metastasis

Surgery:

* See Disease Characteristics
* At least 14 days since prior major surgery and recovered

Other:

* No other prior nonhormonal treatment for metastatic disease
* At least 28 days since prior herbal preparations (e.g., PC-SPES) and recovered
* No other concurrent anticancer medications

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-04

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Carducci, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (8):
- United States (8):
  - Arizona Oncology Associates, Tucson, Arizona
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - Lucille Parker Markey Cancer Center, University of Kentucky, Lexington, Kentucky
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania